CLINICAL TRIAL: NCT01452919
Title: A Phase 3, Short-Term, Multicenter, Placebo-Controlled, Randomized Withdrawal Study of LY2140023 Monohydrate in Patients With DSM-IV-TR Schizophrenia
Brief Title: A Physical Dependence Study in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14326; H8Y-MC-HBDF (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
Keywords: schizophrenia, LY2140023, pomaglumetad methionil
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; pomaglumetad methionil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2140023/LY2140023 (Experimental): Open label phase: 40 milligram (mg) LY2140023 administered orally; given twice daily for up to 4 weeks. At the discretion of the investigator, dose may be adjusted one time to 80 mg. 80 mg dose may be adjusted back to 40 mg one time. Current dose level at randomization will remain constant through the double blind phase.
  Double blind phase: 40 mg or 80 mg LY2140023 administered orally; given twice daily for up to 3 weeks.
  Interventions: Drug: LY2140023
- LY2140023/Placebo (Placebo Comparator): Open label phase: 40 mg LY2140023 administered orally; given twice daily for up to 4 weeks. At the discretion of the investigator, dose may be adjusted one time to 80 mg. 80 mg dose may be adjusted back to 40 mg one time.
  Double blind phase: placebo administered orally; given twice daily for up to 3 weeks.
  Interventions: Drug: LY2140023; Drug: Placebo

INTERVENTIONS:
Drug: LY2140023 — Administered orally
  Other Names: pomaglumetad methionil
Drug: Placebo — Administered orally
  Arms: LY2140023/Placebo

SUMMARY:
The purpose of this study is to determine whether or not people with schizophrenia who take LY2140023 become physically dependent on it, and experience a series of symptoms such as craving to have the drug when they stop using it.

This trial consists of two phases: An open-label phase consisting of up to 4 weeks and a double-blind phase consisting of up to 3 weeks.

DETAILED DESCRIPTION:
This was a short-term, multicenter, placebo-controlled, randomized withdrawal study comparing LY2140023 with placebo in the treatment of outpatients with Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR [APA 2000]) schizophrenia. Patients were male or female outpatients, 18 to 65 years of age (inclusive) at study entry, with a diagnosis of schizophrenia as defined in the DSM-IV-TR

The primary objective of this study was to assess whether LY2140023, when administered in an acute-treatment trial with flexible doses (40 mg or 80 mg) BID, was associated with physical dependence, as measured by the occurrence of withdrawal symptoms during a randomized withdrawal phase in patients diagnosed with schizophrenia. Assessment was to be based on a comparison of randomized LY2140023-treated patients with those on placebo, as measured by the maximum of the 3-day moving average of the patient's total score on the Discontinuation Symptom Checklist-Modified Rickels (DSCMR).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Female participants of childbearing potential must test negative for pregnancy at study entry and agree to use a single, effective, medically acceptable method of birth control
* Participants must require a modification of antipsychotic medication or the initiation of antipsychotic medication, as indicated by their present clinical psychiatric status and/or treatment tolerability as outpatients
* Participants must be considered reliable and have a level of understanding sufficient to perform all tests and examinations required, and be willing to perform all study procedures
* Participants must be able to understand the nature of the study and have given their own informed consent

Exclusion Criteria:

* Have a Clinical Global Impression-Severity Scale (CGI-S) score >4 at study entry
* Have any other psychiatric diagnoses in addition to schizophrenia
* Participants who have a history of inadequate clinical response to antipsychotic treatment for schizophrenia
* Participants who have received an adequate treatment trial, in the opinion of the investigator, with clozapine at doses >200 mg daily within 12 months prior to study entry, or who have received any clozapine at all during the month before study entry
* Participants who are actively suicidal
* Female participants who are pregnant, nursing, or who intend to become pregnant within 30 days of completing the study
* Have known, uncorrected, narrow-angle glaucoma
* Participants who have had electroconvulsive therapy (ECT) within 3 months of study entry or who will have ECT at any time during the study
* Participants with known medical history of human immunodeficiency virus positive (HIV+) status
* Participants who test positive for Hepatitis C virus antibody or Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody
* Participants with current or a history of seizure disorder, uncontrolled diabetes, certain diseases of the liver, renal insufficiency, uncontrolled thyroid condition or other serious or unstable illnesses
* Participants with a corrected QT interval (Bazett's; QTcB) >450 milliseconds (msec) (male) or >470 msec (female) at study entry (based on the central vendor's electrocardiogram [ECG] overread)
* Have previously completed or withdrawn from this study, or any other study investigating LY2140023 or any predecessor molecules with glutamatergic activity
* Are currently enrolled in, or discontinued within the last 60 days from, a clinical trial involving an investigational product for unapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chaïdári, Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tripoli

REFERENCES:
- [Derived] Stauffer VL, Baygani SK, Kinon BJ, Krikke-Workel JO. A short-term, multicenter, placebo-controlled, randomized withdrawal study of a metabotropic glutamate 2/3 receptor agonist using an electronic patient-reported outcome device in patients with schizophrenia. J Clin Psychopharmacol. 2014 Oct;34(5):552-8. doi: 10.1097/JCP.0000000000000187. PMID 25006819

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 4-week open-label treatment period and a 2-week double-blind randomized withdrawal treatment period.
Groups:
- LY2140023 (Open-Label ): 40 milligram (mg) or 80 mg LY2140023 administered orally, twice daily for 4 weeks during open-label treatment period.
- Placebo (Randomization): Placebo administered orally, twice daily for 2 weeks during double-blind, randomized withdrawal treatment period.
- LY2140023 (Randomization): 40 mg or 80 mg LY2140023 administered orally, twice daily for 2 weeks during double-blind, randomized withdrawal treatment period.
Period: Open-Label Treatment
Arm/Group | LY2140023 (Open-Label ) | Placebo (Randomization) | LY2140023 (Randomization)
Started | 123 (During the open label treatment, all patients received LY2140023 monotherapy (first column); no patients were randomized yet (thus, 0 patients listed in column 2 and 3)) | 0 | 0
Received at Least 1 Dose of Study Drug | 123 | 0 | 0
Completed | 103 | 0 | 0
Not Completed | 20 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Perceived lack of efficacy | 3 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Subject is moving or has moved | 1 | 0 | 0
Period: Randomization Treatment
Arm/Group | LY2140023 (Open-Label ) | Placebo (Randomization) | LY2140023 (Randomization)
Started | 0 | 50 (For randomization treatment, the 103 completers of the open label period above were assigned to placebo (50 patients; column 2) and LY2140023 (randomization) (53 patients) (column 3)) | 53 (For randomization treatment, the 103 completers of the open label period above were assigned to placebo (50 patients; column 2) and LY2140023 (randomization) (53 patients) (column 3))
Received at Least 1 Dose of Study Drug | 0 | 50 | 53
Completed | 0 | 47 | 51
Not Completed | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Subject is moving or has moved | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: 40 milligram (mg) or 80 mg LY2140023 administered orally, twice daily for 4 weeks during open-label treatment period.
  Placebo, or 40 mg or 80 mg LY2140023 administered orally, twice daily for 2 weeks during double-blind, randomized withdrawal treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.86 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 118
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 82
  White | 35
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 107
  Greece | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum 3-Day Moving Average (MA) of the Discontinuation Symptom Checklist-Modified Rickels Total Score
Description: The checklist is a 30-item, participant-rated scale that asks whether participants experience symptoms such as nausea, vomiting, loss of appetite, anxiety, irritability, or craving for study drug during the previous day to assess potential symptoms of drug withdrawal. Each item is rated on a 0 (not at all) to 3 (severe). Total scores range from 0-90. Higher scores indicate greater severity of symptoms. The 3-day MA was calculated starting the third day until the last day of double-blind, randomized period. The 3-day MA was the average of scores from that day and previous 2 days. If scores from any of the days during the 3-day was missing, the average was based on the non-missing days. If there was no total scores for any day of the 3-day, the average was considered to be missing. An analysis of covariance (ANCOVA) was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline total score, treatment, pooled investigative site and gender.
Time Frame: Randomization up to Week 2 of randomization treatment
Population: All randomized participants who received at least one dose of study drug and had Discontinuation Symptom Checklist-Modified Rickels total score measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 52
units on a scale | 13.23 (0.96) | 11.50 (0.99)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.170, Type 3 sums of squares — Two-sided p-value; LS Mean Differences = -1.73, Standard Error of Mean 1.25

2. Secondary Outcome: Change From Randomization up to Week 2 in the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-Ar) Total Score
Description: The CIWA-Ar is a 10-item scale that was used to monitor for symptoms of drug withdrawal. The scale includes the following domains/criteria: nausea, vomiting; anxiety; paroxysmal sweats; tactile disturbances; visual disturbances; tremors; agitation; orientation and clouding of sensorium; auditory disturbances; and headache. Items 1-9 have possible scores of 0 (no symptom)-7 (severe symptom), and item 10 has possible scores of 0 (no symptom)-4 (severe symptom). Total scores range from 0-67. Higher scores indicate greater severity of symptom. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline CIWA-Ar total score, treatment, gender, pooled investigative site, visit, baseline CIWA-Ar total score*visit and treatment*visit.
Time Frame: Randomization, randomization treatment Weeks 0.5 and 1 and 1.5 and 2
Population: All randomized participants who received at least one dose of study drug and had CIWA-Ar measurements at randomization and specified post-randomization visits.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 53
units on a scale
  Week 0.5 | -0.7 (0.3) | 0.0 (0.3)
  Week 1: number analyzed (Participants) | 49 | 52
  Week 1 | -0.9 (0.3) | -0.5 (0.3)
  Week 1.5: number analyzed (Participants) | 47 | 51
  Week 1.5 | -0.8 (0.3) | -0.6 (0.3)
  Week 2: number analyzed (Participants) | 47 | 51
  Week 2 | -0.4 (0.3) | -0.5 (0.3)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.109, Type 3 sums of squares — Two-sided p-value. P-value is for Week 0.5; LS Mean Differences = 0.8, Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.372, Type 3 sums of squares — Two-sided p-value. P-value is for Week 1; LS Mean Differences = 0.4, Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.555, Type 3 sums of squares — Two-sided p-value. P-value is for Week 1.5; LS Mean Differences = 0.2, Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.806, Type 3 sums of squares — Two-sided p-value. P-value is for Week 2; LS Mean Differences = -0.1, Standard Error of Mean 0.4

3. Secondary Outcome: Change From Randomization to Week 2 in Barnes Akathisia Scale (BAS) Global Score
Description: The BAS is a 4-item instrument that evaluates akathisia associated with use of antipsychotic medications. Item 4 is the Global Clinical Assessment (Global Score) and is rated 0 to 5 (0 = absent, 5 = severe). The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline BAS global score, treatment, gender, pooled investigative site, visit, baseline BAS global score*visit and treatment*visit.
Time Frame: Randomization, randomization treatment Week 2
Population: All randomized participants who received at least one dose of study drug and had BAS global score measurement at randomization and at least one post-randomization BAS global score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 53
units on a scale | -0.0 (0.0) | -0.0 (0.0)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.762, Type 3 sums of squares — Two-sided p-value; LS Mean Differences = -0.0, Standard Error of Mean 0.0

4. Secondary Outcome: Change From Randomization to Week 2 in Simpson-Angus Scale (SAS) Total Score
Description: The SAS is used to measure parkinsonian-type symptoms in participants exposed to antipsychotics. SAS consists of 10 items; each rated on a 5-point scale, with 0 meaning complete absence of the condition and 4 meaning the presence of the condition in extreme form. The total score is obtained by adding the ten items, and ranges from 0 to 40. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline SAS total score, treatment, gender, pooled investigative site, visit, baseline SAS total score*visit and treatment*visit.
Time Frame: Randomization, randomization treatment Week 2
Population: All randomized participants who received at least one dose of study drug and had SAS total score measurement at randomization and at least one post-randomization SAS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 53
units on a scale | -0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.506, Type 3 sums of squares — Two-sided p-value; LS Mean Differences = 0.0, Standard Error of Mean 0.1

5. Secondary Outcome: Change From Randomization to Week 2 in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS is a 12-item scale designed to record the occurrence of dyskinetic movements. Items 1 to 10 are rated on a 5- point scale, with 0 being no dyskinetic movements and 4 being severe dyskinetic movements. Items 11 and 12 are yes/no questions regarding the dental condition of a subject. The AIMS 1-7 total score is the total of items 1 through 7 of the AIMS, and ranges from 0 to 28. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline AIMS 1-7 total score, treatment, gender, pooled investigative site, visit, baseline AIMS 1-7 total score*visit and treatment*visit.
Time Frame: Randomization, randomization treatment Week 2
Population: All randomized participants who received at least one dose of study drug and had AIMS total score measurement at randomization and at least one post-randomization AIMS total score.
Measure: Least Squares Mean (Standard Error); unit: units a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 53
units a scale | 0.0 (0.1) | -0.0 (0.1)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.515, Type 3 sums of squares — Two-sided p-value; LS Mean Differences = -0.1, Standard Error of Mean 0.1

6. Secondary Outcome: Percentage of Participants With Suicidal Behaviors and Ideations Measured Using the Columbia Suicide Severity Rating Scale (C-SSRS) During Open-Label Treatment Period
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. The percentage of participants with treatment-emergent suicidal ideation or behavior during open-label treatment period (with a change from baseline in C-SSRS) was calculated as the number of participants with an increase in suicidal behavior or ideation over baseline (before open-label treatment), divided by the total number of participants multiplied by 100.
Time Frame: Baseline up to Week 4 of open-label treatment
Population: All enrolled participants who received at least one dose of study drug and had a baseline (before open-label treatment) and at least one post-baseline (during open-label treatment) C-SSRS measurement.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: 40 milligram (mg) or 80 mg LY2140023 administered orally, twice daily for 4 weeks during open-label treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 122
percentage of participants
  Treatment-Emergent Suicidal Ideation | 1.6
  Treatment-Emergent Suicidal Behavior | 0.0

7. Secondary Outcome: Percentage of Participants With Suicidal Behaviors and Ideations Measured Using the Columbia Suicide Severity Rating Scale (C-SSRS) During Double-Blind Randomized Treatment Period
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. The percentage of participants with treatment-emergent suicidal ideation or behavior during double-blind randomized treatment period (with a change from baseline in C-SSRS) was calculated as the number of participants with an increase in suicidal behavior or ideation over baseline (randomization), divided by the total number of participants multiplied by 100.
Time Frame: Randomization up to Week 2 of randomization treatment
Population: All participants who received at least one dose of study drug and had C-SSRS measurement at randomization and at least one post-randomization C-SSRS measurement.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (Randomization): Placebo administered orally, twice daily for 2 weeks during double-blind randomized withdrawal treatment period.
- LY2140023 (Randomization): 40 mg or 80 mg LY2140023 administered orally, twice daily for 2 weeks during double-blind randomized withdrawal treatment period.
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 53
percentage of participants
  Treatment-Emergent Suicidal Ideation | 0.0 | 0.0
  Treatment-Emergent Suicidal Behavior | 0.0 | 0.0

8. Secondary Outcome: Change From Randomization to Week 2 in Clinical Global Impression-Severity Scale (CGI-S)
Description: The CGI-S instrument is used to record the severity of mental illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline CGI-S score, treatment, gender, pooled investigative site, visit, baseline CGI-S score*visit and treatment*visit.
Time Frame: Randomization, randomization treatment Week 2
Population: All randomized participants who received at least one dose of study drug and had CGI-S measurement at randomization and at least one post-randomization CGI-S measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 50 | 53
units on a scale | -0.2 (0.1) | -0.0 (0.1)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.966, Type 3 sums of squares — One-sided p-value; LS Mean Differences = 0.2, Standard Error of Mean 0.1

9. Secondary Outcome: Change From Randomization to Week 2 in Brief Psychiatric Rating Scale (BPRS) Total Scores
Description: BPRS is an 18-item clinician-administered scale used to assess the degree of severity of a participant's general psychopathological symptoms. Item scores range from 1 (not present) to 7 (extremely severe). Total Scores range from 18 to 126. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measure (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values are controlled for baseline BPRS total score, treatment, gender, pooled investigative site, visit, baseline BPRS total score*visit and treatment*visit.
Time Frame: Randomization, randomization treatment Week 2
Population: All randomized participants who received at least one dose of study drug and had BPRS total score measurement at randomization and at least one post-randomization BPRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Randomization) | LY2140023 (Randomization)
Number analyzed (Participants) | 49 | 52
units on a scale | -2.20 (0.55) | -1.28 (0.54)
Statistical Analysis 1: Comparison: Placebo (Randomization) vs LY2140023 (Randomization); Test type: Superiority or Other; p = 0.895, Type 3 sums of squares — One-sided p-value; LS Mean Differences = 0.92, Standard Error of Mean 0.73

ADVERSE EVENTS:
Arm/Group | LY2140023 (Open-Label ) | Placebo (Randomization) | LY2140023 (Randomization)
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/50 | 0/53
Other Adverse Events (participants affected / at risk) | 83/123 | 13/50 | 20/53
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2140023 (Open-Label ) (N=123) | Placebo (Randomization) (N=50) | LY2140023 (Randomization) (N=53)
Hearing impaired (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 35 (39) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (17) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 9 (9) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 19 (20) | 4 (4) | 1 (2)
Somnolence (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 10 (12) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 8 (9) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 10 (11) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days